CLINICAL TRIAL: NCT04499599
Title: Randomized, Single-blinded, Controlled, Parallel-arm Study to Evaluate the Effect of Fast Bar(TM) on Physiological Fasting Condition
Brief Title: Effects of Fast Bar on Physiological Fasting
Acronym: FastBar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L-Nutra Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20201920
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Fasting
Keywords: Fast Bar; Fasting; Intermittent fasting; Ketone bodies; ß-hydroxybutyrate
MeSH Terms: conditions — Fasting; Intermittent Fasting | interventions — Meals; Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: For comparison between the placebo breakfast bar and the Fast Bar groups, the participants are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fast Group (Active Comparator): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 19 hours.
  Interventions: Other: Dinner; Other: Fasting
- Breakfast Group (Placebo Comparator): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 15 hours and then consume a breakfast bar on day 2.
  Interventions: Other: Dinner; Other: Fasting; Other: Study food
- Fast Bar Group (Experimental): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 15 hours and then consume a Fast Bar on day 2.
  Interventions: Other: Dinner; Other: Fasting; Other: Study food

INTERVENTIONS:
Other: Dinner — Study subjects will consume a standardized ready-to-eat meal as dinner.
Other: Fasting — Subjects in all groups will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1 and then fast overnight for approximately 15 hours.
Other: Study food — Study subjects will either continue to fast for 6 hours (Fast Group), consume either a breakfast (Breakfast Group) or a Fast Bar (Fast Bar Group).
  Arms: Breakfast Group; Fast Bar Group

SUMMARY:
This study evaluates how Fast Bar(TM), a specially formulated energy bar, affects the physiological condition in participants after an overnight fasting. Participants will fast for 19 hours (Fast Group), consume a breakfast Bar (Breakfast Group) or a Fast Bar(TM) (Fast Bar Group) after an approximately 15-hour overnight fasting. Participants will be assessed for physiological parameters associated with fasting.

DETAILED DESCRIPTION:
Interest in fasting-based programs (i.e. intermittent fasting) for improvement of health and longevity continues to grow. While benefits of intermittent fasting have been convincingly demonstrated in rodent models, the more limited data in humans is less clear.

The short-term fasting (e.g. 12 to 48 hours in duration) utilized in many intermittent fasting programs are considered safe, but some individuals may find them subjectively difficult. As such, the question of whether the benefits of fasting can be obtained while small amounts of food are consumed is of substantial interest.

One commercially available product that is designed to be consumed during periods of intermittent fasting is the Fast Bar™,which stems out of the well-researched fasting-mimicking diet to assist prolonged fasting. The unique formulation of the Fast Bar™ is hypothesized to minimize deviations in metabolic biomarkers associated with a fasting state. This may allow for extension of a fasting period through reduced subjective difficulty of fasting.The objective of this study is to evaluate the metabolic and subjective effects of consuming a novel food product (Fast Bar™) after a short period of fasting.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent;
* Ability and willingness to use Zoom teleconference;
* Ability and willingness to perform the study tests and adhere to study protocol (to the best of the participant's knowledge);
* BMI 20-35 kg/m2 (inclusive) at screening;
* In good health (as determined by medical history to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days).

Exclusion Criteria:

* Has any medical disease or condition that, in the opinion of the principal investigator (PI) or appropriate study personnel, precludes study participation* (*Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial);
* History of gastric bypass (based on medical history provided at screening);
* Under medications aimed at keeping blood glucose under control (based on medical history provided at screening);
* Type 1 diabetes (based on medical history provided at screening);
* Taking insulin, insulin analogs, or octreotide (based on medical history provided at screening);
* Food allergies which would make the subject unable to consume the food provided (based on medical history and information provided at screening) (participants will be asked to review the ingredient lists for the dinner meal, the breakfast and the Fast Bar, and to state that they are not allergic to the ingredients to the best of their knowledge);
* Women who are pregnant;
* Alcohol dependency (alcohol intake greater than two drinks per day for women and three drinks per day for men) (based on medical history and information provided at screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Hsu, MD, Principal Investigator — L-Nutra Inc
Locations (1):
- L-Nutra Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fast Group | Breakfast Group | Fast Bar Group
Started | 35 | 35 | 35
Completed | 35 | 35 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fast Group | Breakfast Group | Fast Bar Group | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.5) | 45.9 (12.5) | 46.4 (10.9) | 46.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 23 | 72
  Male | 8 | 13 | 12 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 27 | 30 | 82
  Black | 2 | 3 | 1 | 6
  Hispanic | 7 | 2 | 3 | 12
  Asian | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Ketone Area Under the Curve
Description: Blood ketone (ß-hydroxybutyrate, BHB) area under the curve (AUC) will be measured with a Abbott Precision Xtra Blood Glucose and Ketone Monitoring Meter Kit on 0, 1, 2, 3, and 4 hours after consuming the study foods.
Time Frame: BHB Area Under the Curve between 0 to 4 hours after consuming the study foods
Measure: Mean (Standard Deviation); unit: mg/dL*h
Arm/Group | Fast Group | Breakfast Group | Fast Bar Group
Number analyzed (Participants) | 35 | 35 | 35
mg/dL*h | 1.27 (0.53) | 0.62 (0.18) | 1.17 (0.34)

2. Primary Outcome: Glucose Area Under the Curve
Description: Blood glucose area under the curve (AUC) will be measured with a Abbott Precision Xtra Blood Glucose and Ketone Monitoring Meter Kit on 0, 1, 2, 3, and 4 hours after consuming the study foods.
Time Frame: Glucose Area Under the Curve between 0 to 4 hours after consuming the study foods
Measure: Mean (Standard Deviation); unit: mg/dL*h
Arm/Group | Fast Group | Breakfast Group | Fast Bar Group
Number analyzed (Participants) | 35 | 35 | 35
mg/dL*h | 365 (50) | 401.4 (42.3) | 363.5 (37.3)

ADVERSE EVENTS:
Time Frame: 2 days.
Arm/Group | Fast Group | Breakfast Group | Fast Bar Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT04499599/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT04499599/ICF_001.pdf